CLINICAL TRIAL: NCT05835193
Title: Visual Acuity Assessment in Pre-school Students.
Brief Title: Pre-symptomatic Screening of Visual Acuity in Pre-school Students
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: DUTH/EHDE2/20-10-2022
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Visual Acuity; Refractive Errors; Low Vision; Vision Disorders
Keywords: kindergarten; distance visual acuity; pre-school students; reading capacity
MeSH Terms: conditions — Refractive Errors; Vision, Low; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Pre-school students in Alexandroupolis, Greece
  Interventions: Other: Diagnostic Test: Distance Visual Acuity Examination

INTERVENTIONS:
Other: Diagnostic Test: Distance Visual Acuity Examination — Best spectacle-corrected distance visual acuity and reading capacity of pre-school students in Alexandroupolis, Greece will be examined via a web-based digital visual acuity chart

SUMMARY:
The present research process is a prospective, non-interventional clinical study that will be conducted -under the auspices of the Democritus University of Thrace (DUTH)- in the pre-school students of the city of Alexandroupolis, Greece.

* The study aims to assess the visual acuity of the kindergarten students.
* The measurement of monocular best-spectacle corrected visual acuity will be performed using a web-based visual acuity chart

DETAILED DESCRIPTION:
Study protocol will adhere to the tenets of the Declaration of Helsinki and written informed consent will be obtained by the legal guardians of all participants.

The measurement of the visual acuity (monocular and binocular) will be performed using DDART, a digital visual acuity tool that has been developed and validated by the Democritus University of Thrace and is also an approved Category 1 Medical Device by the country's National Organization for Medicines, via a web-based digital chart in a high-resolution screen. The same environmental lighting conditions and the same screen brightness will be applied. The examination will be performed at the same predetermined viewing distance.

Finally, according to each participant's visual acuity, appropriate instructions will be given for further examinations directly to the legal guardians in order to comply with the GDPR.

ELIGIBILITY:
Inclusion Criteria:

* Pre-school students aged 5-7 years old.

Exclusion Criteria:

* Age >7 years old
* Students with health conditions that do not allow the evaluation of the visual acuity .

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pre-school students aged 5-7 years old
Sampling Method: Non-Probability Sample
Enrollment: 1098 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Best spectacle-corrected distance visual acuity | 1 week
  Visual acuity of each eye using spectacle correction

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece